CLINICAL TRIAL: NCT00395252
Title: Multicenter Phase II-trial to Investigate Safety and Efficacy of an Adjuvant Therapy With Gemcitabine and Erbitux® in Patients With R0 or R1 Resected Pancreatic Cancer
Brief Title: Safety and Efficacy Therapy of Gemcitabine and Erbitux® to R0 or R1 Resected Pancreatic Cancer
Acronym: ATIP
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Carmen Schade-Brittinger (Other)
Responsible Party: Sponsor-Investigator, Carmen Schade-Brittinger, Philipps University, Philipps University Marburg
Organization: Philipps University Marburg (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EUDRACT-No. 2005-005168-94
Record Dates: First submitted 2006-11-01; First posted 2006-11-02 (Estimated); Last update posted 2015-10-02 (Estimated); Status verified 2015-10

CONDITIONS: Adenocarcinoma
Keywords: pancreatic cancer; adjuvant chemotherapy; phase 2; R0 or R1 resected Adenocarcinoma of the Pancreas
MeSH Terms: conditions — Adenocarcinoma; Pancreatic Neoplasms | interventions — Cetuximab; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- one arm study (Experimental): Cetuximab (Erbitux®) and Gemcitabine treatment over 6 months
  Interventions: Drug: Cetuximab (Erbitux®) and Gemcitabine

INTERVENTIONS:
Drug: Cetuximab (Erbitux®) and Gemcitabine — Cetuximab:
  Loading dose of 400 mg/m2, followed by weekly doses of 250 mg/m2. Cetuximab will be administered once weekly for up to 6 months (treatment duration: 24 weeks)
  Gemcitabine:
  1000 mg/m2 administered on days 1, 8, 15 Cycles will be repeated on day 29, up to 6 treatment cycles will be administered
  Mode of administration:
  Intravenous infusion
  Other Names: Cetuximab; Gemzar

SUMMARY:
This is an open-label, non-randomized Phase II study to evaluate immunochemotherapy in patients with R0 OR R1-resected pancreatic cancer.

DETAILED DESCRIPTION:
Available study data indicated a possible benefit from adjuvant chemotherapy for patients with resected pancreatic cancer. The optimal therapy regimen has yet to be determined.

Based on the experiences with cetuximab (Erbitux®)and gemcitabine in advanced pancreatic cancer and with gemcitabine as adjuvant therapy, the aim of this study was to evaluate the feasibility of the combined treatment of cetuximab and gemcitabine in patients with R0 or R1-resectable pancreatic cancer and to evaluate if the disease free survival can be increased by the addition of an EGFR-targeted therapy.

ELIGIBILITY:
Inclusion Criteria:

* Provided signed written informed consent.
* Men and woman age > 18 years
* Histologically confirmed R0 OR R1 resected ductal adenocarcinoma of the pancreas
* Life expectancy >12 weeks
* Patients with performance status of ECOG ≤ 2
* Patients without metastasis

Exclusion Criteria:

* Women of child bearing potential (WOCP) who are unwilling or unable to use an acceptable method to avoid pregnancy for the entire study period and follow-up to 4 weeks after the study.
* Women who are pregnant or breastfeeding.
* Women with a positive pregnancy test on enrollment or prior to study drug administration.
* Dementia, altered mental status, or any psychiatric condition that would prohibit the understanding or rendering of informed consent.
* Any concurrent malignancy other than non-melanoma skin cancer, or carcinoma in situ of the cervix. (Patients with a previous malignancy but without evidence of disease for > 5 years will be allowed to enter the trial).
* Inadequate hematologic function defined by an absolute neutrophils count (ANC) < 1,500/mm³, a platelet count < 100,000/mm³ and a hemoglobin < 9 g/dL.
* Inadequate hepatic function defined by the upper limit of normal (ULN), AST and ALT levels > 5 times the ULN.
* Serum bilirubin > 1.5 times the ULN.
* Inadequate renal function defined by a serum creatinine > 1.5 times the ULN.
* Prior cetuximab or other therapy that targets the EGF pathway.
* Prior antibody therapy.
* Any known allergic reaction against cetuximab.
* Any concurrent chronic systemic immune therapy, radiation therapy, hormonal therapy (except for physiological replacement), or any other investigational agents.
* HIV infection.
* Having participated in another clinical trial in the preceding 30 days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2006-10; Primary Completion 2010-11 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
disease free survival | 18 months after registration

SECONDARY OUTCOMES:
Overall survival
Quality of life
Incidence of Adverse Events | 19 months since registration

CONTACTS AND LOCATIONS:
Overall Officials: Thomas M Gress, Prof.Dr. med, Principal Investigator — Klinik für Gastroenterologie, Endokrinologie und Stoffwechsel, University of Marburg
Locations (8):
- Germany (8):
  - Interdisziplinäres Tumorzentrum (Comprehensive Cancer Center), Fulda
  - Nationales Centrum für Tumorerkrankungen (NCT), Universitätsklinikum Heidelberg, Heidelberg
  - Klinik für Innere Medizin II, Klinikum der Universität Jena, Jena
  - Allgemein-, Viszeral- und Thoraxchirurgie, Klinikum Kassel, Kassel
  - Abt. für Chirurgie, Universitätsklinikum Mannheim gGmbH, Mannheim
  - Klinikum Giessen und Marburg, Standort Marburg, Marburg
  - II Medizinische Klinik und Poliklinik, Klinikum rechts der Isar, TU München, Munich
  - Klinik- und Poliklinik für Innere Medizin I, Klinikum der Universität Regensburg, Regensburg

REFERENCES:
- [Result] Fensterer H, Schade-Brittinger C, Muller HH, Tebbe S, Fass J, Lindig U, Settmacher U, Schmidt WE, Marten A, Ebert MP, Kornmann M, Hofheinz R, Endlicher E, Brendel C, Barth PJ, Bartsch DK, Michl P, Gress TM; Arbeitsgemeinschaft Internistische Onkologie (AIO). Multicenter phase II trial to investigate safety and efficacy of gemcitabine combined with cetuximab as adjuvant therapy in pancreatic cancer (ATIP). Ann Oncol. 2013 Oct;24(10):2576-2581. doi: 10.1093/annonc/mdt270. Epub 2013 Jul 29. PMID 23897705